CLINICAL TRIAL: NCT05877833
Title: An Open-Label, Single-Center, Prospective, Observational, Clinical Use Study Evaluating the Safety and Performance Characteristics of Ephemeral® Tattoo Ink in Healthy Subjects
Brief Title: Evaluating the Safety and Performance Characteristics of Ephemeral® Tattoo Ink in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Ephemeral Solutions Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPHEM-001
Record Dates: First submitted 2023-03-07; First posted 2023-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Tattoo; Pigmentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vibrancy: Healthy adults
  Interventions: Other: Vibrancy Assessment

INTERVENTIONS:
Other: Vibrancy Assessment — Additionally, important medical events that may not result in death, be life threatening, or require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

SUMMARY:
An Open-Label, Single-Center, Prospective, Observational, Clinical Use Study Evaluating the Safety and Performance Characteristics of Ephemeral® Tattoo Ink in Healthy Subjects

DETAILED DESCRIPTION:
Study product will be applied at the baseline visit by a skilled tattoo artist. The tattoo design will be approximately 2 inches x 2 inches and will consist of line work. No filling or shading will be included in the design.

ELIGIBILITY:
Inclusion Criteria:

* ● Subjects who are able to give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA authorization.

  * Healthy adults between 18 and 60 years of age.
  * Subjects with Fitzpatrick photo skin types I-VI.
  * Subjects who agree not to have any procedures affecting skin quality of the arm (Ex. Other tattoo within 2 inches of border of investigational ink, microdermabrasion, acne treatments, hair removal) for the duration of the study.
  * Subjects who understand this study and are able to follow study instructions and are willing to attend the required study visits.
  * Subjects who agree to be photographed for research reasons and their identity may not be concealed in these photographs.
  * Subjects who are willing not to publicize their EPHEMERAL® TATTOO on social media or through any web platform.

Exclusion Criteria:

* ● Subjects who are pregnant, planning to become pregnant or breastfeeding within 16 weeks of participation.

  * Subjects of childbearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy or bilateral oophorectomy.
  * Subjects who cannot understand or are not willing to comply with the requirements of the study.
  * Subjects who have had any procedures affecting skin quality of the arm (Ex. Other tattoo within 2 inches of border of investigational ink, microdermabrasion, acne treatments, hair removal) in the 4 months prior to enrollment.
  * Subjects who have had recent extreme sun exposure to the treatment area (as defined by investigator)
  * Subjects who do not agree to avoid using tanning beds or intensive exposure to the sun for the duration of the study and within two weeks of initiating participation.
  * Subjects who have any dermatologic conditions including acne, rosacea, eczema, psoriasis, actinic keratosis, severe sun damage, infection or scars within the treatment area.
  * Subjects who have an active inflammatory process (skin eruptions such as cysts, pimples, rashes or hives) or infection within the treatment area.
  * Subjects currently taking, or with plans to start, any medication or supplement that may affect clotting, increase risk of infection or cause increased bleeding (Ex: Humira, fish oil, ginseng, aspirin, heparin, warfarin, recent inoculation/flu shot), to be determined by investigator.
  * Subjects who have any known cancer including skin cancers (basal cell carcinoma, squamous cell carcinoma and melanoma) in the treatment area.
  * Subjects who have an existing medical condition that the Investigator considers may put the subject at risk or compromise their participation in the study.
  * Subjects who have participated in another research study in the past 30 days.
  * Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Adults
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with tattoo vibrancy of 50% or greater | 3 months
  To confirm that EPHEMERAL® TATTOO Ink formulation 1 and formulation 2 are able to meet and maintain vibrancy of 50% during the first 3 months after tattoo is applied

SECONDARY OUTCOMES:
To evaluate the degree of healing of EPHEMERAL® TATTOO Ink | 3 months
  To evaluate the degree of healing of EPHEMERAL® TATTOO Ink as measured by the Investigator post-application healing assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Brennal Pierre, Milford, Connecticut, United States